CLINICAL TRIAL: NCT00810498
Title: Comparing Known Modes of Ventilation Delivered by Trilogy Versus Conventional Mechanical Ventilators
Brief Title: Trilogy Comparison Study - Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MR-0609-TRI2-SS
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Insufficiency; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Trilogy (Experimental): Trilogy Device
  Interventions: Device: Trilogy
- Standard of Care (Active Comparator): Participants prescribed ventilator
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Trilogy — Exposure for one hour on the Trilogy ventilator
  Arms: Trilogy
Device: Standard of Care — Exposure to participants current ventilator
  Arms: Standard of Care

SUMMARY:
The objective of this study (Part II) will be to compare the performance of the Trilogy device and a conventional ventilator (participant's current device). Both devices will be set to the participants' current mode and prescription settings.

DETAILED DESCRIPTION:
A. Primary Hypothesis and end-point In patients with respiratory insufficiency, when compared to conventional ventilators, the Trilogy device achieves comparable level of gas exchange (measured as partial pressure of CO2 in arterial or venous blood)and SpO2 levels during various modes of ventilation.

B. Secondary Hypothesis and end-points In patients with respiratory insufficiency, when compared to conventional ventilators, the Trilogy device achieves comparable breathing pattern (tidal volume, respiratory rate, minute ventilation), hemodynamics (heart rate), and subjective measures of breathing comfort (measured by modified Borg dyspnea scale).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years of age; < 85 years of age
2. Able to follow instructions
3. Able to provide informed consent
4. Considered clinically stable, with low flow oxygen requirements less than 15 LPM (or FIO2 less than 60 %) and PEEP no greater than 10 cm H2O.
5. Requiring mechanical ventilation through nasal/facial mask,tracheostomy or endotracheal tube (ET Tube)

Exclusion Criteria:

1. Clinically unstable, i.e.,

   1. Acute Respiratory Failure
   2. Participants with refractory hypotension defined as systolic blood pressure less than 90 mm Hg despite inotropic agents),
   3. Uncontrolled cardiac ischemia or arrhythmias,
   4. or as otherwise determined inappropriate for the study as determined by the investigator.
2. Patients suffering from metastatic or terminal cancer and patients with do-not-resuscitate orders
3. Pregnancy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-03-12 (Actual); Primary Completion 2009-02-05 (Actual); Study Completion 2009-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Mink, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Trilogy First, Then Standard of Care: These participants used Trilogy first, then Standard of Care.
- Standard of Care First, Then Trilogy: these participants used Standard of Care first, then Trilogy.
Period: Overall Study
Arm/Group | Trilogy First, Then Standard of Care | Standard of Care First, Then Trilogy
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Consented: All participants that were consented.
Arm/Group | All Participants Consented
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  Canada | 11

OUTCOME MEASURES:

1. Primary Outcome: Comparable Level of Gas Exchange (Measured as Partial Pressure of CO2 in Arterial or Venous Blood).
Description: Blood gas was obtained for this study one hour after use of each device.
Time Frame: After one hour of ventilator use
Population: Only 10 out of 11 total participants' data were used for blood gases due to one participant's venous line occluding.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Trilogy | Standard of Care
Number analyzed (Participants) | 10 | 10
mm Hg | 42 (14) | 43 (14)

2. Primary Outcome: Comparable Level of Gas Exchange SpO2 Levels During Various Modes of Ventilation.
Description: Pulse Oximetry was measured after one hour of use of each ventilator.
Time Frame: After one hour of ventilator use
Population: Only 10 out of the 11 total participants' data were used for SpO2 due to missing data. Only 8 out of the 11 total participants data were used for SpO2 Standard of care analysis due to missing data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Trilogy | Standard of Care
Number analyzed (Participants) | 10 | 8
mm Hg | 98 (2) | 97 (2)

3. Secondary Outcome: Tidal Volume
Description: Tidal volume is the amount of air that moves in or out of the lungs with each respiratory cycle. It measures around 500 mL in an average healthy adult male and approximately 400 mL in a healthy female. Average tidal volume was compare after a hour of use of each device.
Time Frame: One hour during ventilator use.
Population: Missing one data set for Standard of care.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Trilogy | Standard of Care
Number analyzed (Participants) | 11 | 10
mL/kg | 479 (182) | 498 (128)

4. Secondary Outcome: Minute Ventilation
Description: Minute ventilation is the volume of gas inhaled or exhaled from a person's lungs per minute. This was measured after one hour of use of each device.
Time Frame: One hour during ventilator use.
Population: Missing one data set for Standard of Care.
Measure: Mean (Standard Deviation); unit: L/m
Arm/Group | Trilogy | Standard of Care
Number analyzed (Participants) | 11 | 10
L/m | 10.11 (1.94) | 10.11 (2.12)

5. Secondary Outcome: Hemodynamics (Heart Rate)
Description: Number of beats per minute. Measured after one hour of use of each device.
Time Frame: One hour during ventilator use.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Trilogy | Standard of Care
Number analyzed (Participants) | 11 | 11
beats per minute | 89.9 (19.0) | 90.4 (19.7)

ADVERSE EVENTS:
Groups:
- Trilogy Device: Trilogy Device
  Trilogy: Exposure for one hour on the Trilogy ventilator
Arm/Group | Trilogy Device | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No